CLINICAL TRIAL: NCT03959761
Title: To Assess the Tolerance of Intraperitoneal (IP) Nivolumab After Extensive Debulking Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients With Advanced Ovarian Carcinoma, Through a Phase Ib/II Study Including Patients at 3 Dose-levels for Nivolumab
Brief Title: Tolerance of Intraperitoneal (IP) Nivolumab After Extensive Debulking Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients With Advanced Ovarian Carcinoma
Acronym: ICONIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0802; 2018-004408-21 (Other: ID-RCB)
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
Keywords: Immunotherapy; Debulking surgery; Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Infusions, Parenteral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Intraperitoneal (IP) nivolumab treatment, after extensive debulking surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
  Interventions: Drug: Intraperitoneal (IP) nivolumab infusion

INTERVENTIONS:
Drug: Intraperitoneal (IP) nivolumab infusion — Patients will be treated according to three dose-levels of nivolumab, starting 5 to 7 days after surgery + Hyperthermic Intraperitoneal Chemotherapy (HIPEC), through an Intraperitoneal (IP) catheter :
  * Level 1 : 0.5 milligrams/kilogram (mg/kg) IP infusion, repeated every 2 weeks for 4 infusions
  * Level 2 : 1 mg/kg IP infusion, repeated every 2 weeks for 4 infusions
  * Level 3 : 3 mg/kg IP infusion, repeated every 2 weeks for 4 infusions
  * Level -1 : 0,3 mg/kg IP infusion, repeated every 2 weeks for 4 infusions

SUMMARY:
Spread pattern, the lack of alternative treatments, and emerging data on the activity of anti-Programmed death ligand 1 (PDL1) targeted checkpoint inhibitor therapy in gynecological cancers provide the rationale for this investigation.

Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) are likely to increase the tumor-antigen expression and the mutational load. As a result, it would be interesting to combine this approach with immunotherapy. Moreover, Intraperitoneal (IP) infusion will directly target the peritoneal cavity and potentially enhance the immune response. Indeed some recent papers indicate that the peritoneum could be considered as a lymphoid organ, involving "milky spots", thus able to produce a better immune response when immunotherapy is given by IP route rather than intravenous (IV) route.

The investigating team in Lyon, France is one of the major groups for HIPEC research in Europe (Pr O. Glehen et al) - Reference center for the tumors of the peritoneum (French National Cancer Institute).

The aim of this study is to assess in this I/II phase study, the feasibility of extensive debulking surgery and HIPEC followed by Intraperitoneal (IP) nivolumab dose escalation in patients with advanced ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Signed informed consent and ability to comply with treatment and follow-up.
* Histological or cytological proven primary epithelial ovarian carcinoma or peritoneal cancer or fallopian tube carcinoma in relapse, including serous papillary adenocarcinoma, mucinous adenocarcinoma, clear-cell carcinoma, undifferentiated carcinoma, mixed mullerian tumor and endometrioid adenocarcinoma. Patients with low grade tumors can be included.
* Not eligible for front-line cytoreduction in first platinum-sensitive relapse
* Eligible for surgical cytoreduction and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) after one or more lines of chemotherapy. All chemotherapy regimens usually recommended for the treatment of ovarian cancer are accepted :

  * Platinum based regimens +/- bevacizumab for the treatment of platinum sensitive disease.
  * Non - platinum based regimens +/- bevacizumab for the treatment of platinum resistant disease.
* Satisfactory haematological evaluation: neutrophil rate greater than 1500/millimeters cubed, platelet count greater than 100 grams/liter;
* Satisfactory renal and hepatic function: serum creatinine ≤1.5 times the normal upper values or creatinine clearance ≥50 milliliters/minute, bilirubin ≤1.25 times upper normal values, ratio aspartate transaminase/alanine transaminase (AST/ALT) ≤1.5 times the upper normal values (≤5 times the upper normal values for patients with liver metastases)
* No unstable conditions: myocardial infarction within 6 months prior to the start of the study, congestive heart failure, unstable angina, active cardiomyopathy, unstable rhythm disorder, uncontrolled hypertension, uncontrolled psychiatric disorders, severe infection, peptic ulcer or any condition that could be aggravated by treatment or limit compliance (investigator assessment)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to the start of study drug.
* Women of childbearing potential should use an adequate method of contraception to avoid pregnancy during nivolumab treatment until 5 months after the last dose of investigational drug.

Exclusion Criteria:

* Ovarian cancer in first-line
* First platinum sensitive relapse amenable to initial cytoreduction surgery
* History of breast cancer or previous malignancies within 5 years prior to inclusion, with the exception of radically excised basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded
* Patients with active coronary artery disease
* Patients with known acute hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive, that might affect host immunity
* Patients with known pre-existent auto-immune disease
* Patients with severe restrictive or obstructive pulmonary disease
* Known carboplatin or cisplatin allergy
* Life expectancy less than 3 months
* Extraperitoneal metastases for which the site or number preclude potentially curative surgery at any moment during the course of the disease
* Sign of bowel obstruction or lesions whose topography indicates a risk of intestinal perforation or inflammatory bowel disease
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 3-4
* Contraindication to the placement of an intraperitoneal catheter
* peripheral sensory neuropathy grade at least 2
* Patient with myelodysplastic syndrome/acute myeloid leukemia history.
* Major surgery within 4 weeks of starting study treatment and patient must have recovered from any effects of any major surgery.
* Previous allogenic bone marrow transplant
* Any previous treatment with Anti programmed cell death 1 (PD-1) immunotherapy
* Pregnant or lactating women
* Unable to give consent
* Patient under legal protection measures
* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Safety profile of the Intraperitoneal (IP) nivolumab treatment | 28 days
  Safety profile of the Intraperitoneal (IP) nivolumab treatment, after extensive debulking surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC), as defined by the maximal dose for which a Dose-Limiting Toxicity (DLT) will be observed in no more than 1 patient out of 6 patients included at the respective dose-level.

SECONDARY OUTCOMES:
Changes over time in disease progression | Measure taken at 1 month, 3 months, 6 months
  Clinical diease progression is defined as the occurence and persistance of symptoms which are considered by the investigator as undoubtfully disease-related. Disease progression will be clinically evaluated using body imaging scans at different times after the last Intraperitoneal (IP) nivolumab injection.
Changes in toxicity as assessed by the Common Terminology Criteria (CTC) scale- Surgery | Measure taken at Day 5, Day 20, Day 35, and Day 50 after Surgery
  The National Cancer Institute created originally the Common Toxicity Criteria (CTC) to aid in the recognition and grading severity of adverse effects caused by chemotherapy treatments. The grading scale is as follows with grade 0 being no cancer and grade 5 being death:
  Grade Description Grade 0 (none) None Grade 1 (mild) Painless ulcers, erythema, or mild soreness in the absence of lesions Grade 2 (moderate) Painful erythema, oedema, or ulcers but eating or swallowing possible Grade 3 (severe) Painful erythema, oedema, or ulcers requiring intravenous (IV) hydration Grade 4 (life-threatening) Severe ulceration or requiring parenteral or enteral nutritional support or prophylactic intubation Grade 5 (death) Death related to toxicity
Changes over time in toxicity as assessed by the Common Terminology Criteria (CTC) scale- Intraperitoneal (IP) nivlumab infusion | Measure taken at 1 month, 3 months and 6 months after the last IP nivlumab infusion
  The National Cancer Institute created originally the Common Toxicity Criteria (CTC) to aid in the recognition and grading severity of adverse effects caused by chemotherapy treatments. The grading scale is as follows with grade 0 being no cancer and grade 5 being death:
  Grade Description Grade 0 (none) None Grade 1 (mild) Painless ulcers, erythema, or mild soreness in the absence of lesions Grade 2 (moderate) Painful erythema, oedema, or ulcers but eating or swallowing possible Grade 3 (severe) Painful erythema, oedema, or ulcers requiring intravenous (IV) hydration Grade 4 (life-threatening) Severe ulceration or requiring parenteral or enteral nutritional support or prophylactic intubation Grade 5 (death) Death related to toxicity
Changes in tolerance of post procedure intravenous (IV) chemotherapy- Surgery | Measure taken at Day 5, Day 20, Day 35, and Day 50 after surgery
  Patients will be clinically evaluated for any changes in tolerance to post procedure intravenous (IV) chemotherapy as defined by the appearance of any serious adverse events.
Changes over time in tolerance of post procedure intravenous (IV) chemotherapy- Intraperitoneal (IP) nivlumab infusion | Measure taken at 1 month, 3 months and 6 months after the last IP nivlumab infusion
  Patients will be clinically evaluated for any changes in tolerance to post procedure intravenous (IV) chemotherapy which includes any serious adverse events at different times after the last IP nivlumab infusion

CONTACTS AND LOCATIONS:
Overall Officials: Gilles FREYER, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Corbaux P, Freyer G, Glehen O, You B, Bakrin N, Gelot A, Dayde D, Sajous C, Piffoux M, Peron J, Lescuyer G, Payen L, Kepenekian V. Intraperitoneal Nivolumab after Debulking Surgery and Hyperthermic Intraperitoneal Chemotherapy in Advanced Ovarian Cancer: A Phase I Study with Expansion Cohort. Clin Cancer Res. 2024 Aug 15;30(16):3438-3446. doi: 10.1158/1078-0432.CCR-24-0507. PMID 38819408